CLINICAL TRIAL: NCT01477385
Title: Treatment of Initial Caries Lesions on Proximal Surfaces of Primary and Permanent Posterior Teeth: a Randomized Placebo-controlled Study.
Brief Title: Treatment of Initial Caries Lesions on Proximal Surfaces of Primary and Permanent Posterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mariana Minatel Braga, Phd, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDFtrials-01
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Dental Caries; Compliance Behavior
Keywords: dental caries; primary teeth; permanent teeth; silver diamine fluoride
MeSH Terms: conditions — Dental Caries; Patient Compliance | interventions — icon infiltrant; silver diamine fluoride; Dental Devices, Home Care; Oral Hygiene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resin Infiltration (Active Comparator): Resin Infiltration 30% Silver Diammine Fluoride Placebo Dental Flossing
  Interventions: Procedure: Resin Infiltration; Procedure: Dental Flossing; Procedure: 30% Silver Diammine Fluoride Placebo
- 30% Silver Diammine Fluoride (Experimental): 30% Silver Diammine Fluoride Resin Infiltration Placebo Dental Flossing
  Interventions: Procedure: 30% Silver Diammine Fluoride; Procedure: Dental Flossing; Procedure: Resin Infiltration Placebo
- Oral Hygiene (Active Comparator): Dental Flossing 30% Silver Diammine Fluoride Placebo Resin Infiltration Placebo
  Interventions: Procedure: Dental Flossing; Procedure: Resin Infiltration Placebo; Procedure: 30% Silver Diammine Fluoride Placebo

INTERVENTIONS:
Procedure: Resin Infiltration — After cleaning the proximal surface with caries lesion, it will be performed the local infiltration anesthesia and adaptation of the rubber dam. The adjacent tooth will be protected by plastic or metal strip. Hydrochloric acid 15% will be applied on the lesion, which will be washed and dried. The surface should be dried by applying 95% ethanol and air-way syringe. The resin infiltration (Icon, DMG) will be applied on the lesion. The resin will be polymerized and applied again and polymerized.
  Other Names: Icon
  Arms: Resin Infiltration
Procedure: 30% Silver Diammine Fluoride — It will be cleaned like group I. Soft tissues will be protected with petroleum jelly. The 30% silver diamine fluoride (Cariestop, Biodinamica) will be applied with a disposable microbrush for 3m. Then the surface will be washed for 30s.
  Other Names: Cariestop
  Arms: 30% Silver Diammine Fluoride
Procedure: Dental Flossing — In this group, the patient will perform only mechanical removal of biofilm to floss daily.
  Other Names: Oral hygiene
Procedure: Resin Infiltration Placebo — In this group, the patient will be held only inserting the rubber dam and applied sterile water as a substitute for acid, ethanol and resin infiltration.
  Other Names: Icon Placebo
  Arms: 30% Silver Diammine Fluoride; Oral Hygiene
Procedure: 30% Silver Diammine Fluoride Placebo — Soft tissues will be protected with petroleum jelly. The patient will receive sterile water application with a disposable microbrush for 3m. Then the surface will be washed for 30s.
  Other Names: Cariestop Placebo
  Arms: Oral Hygiene; Resin Infiltration

SUMMARY:
This study aims to evaluate the effectiveness of 30% silver diamine fluoride in the treatment of clinically caries lesions in enamel, with radiographic image restricted to the enamel or the outer third of dentin on the proximal surfaces of primary and permanent posterior teeth. It also aims to compare it to the resin infiltration and to the control of proximal biofilm through the oral hygiene.

DETAILED DESCRIPTION:
The sample will be comprised of 141 patients between 3 to 10 year-old and 504 proximal surfaces of 12-to-17-year-old adolescents, who present at least one proximal surface with initial caries lesion. Patients will be randomly allocated to treatments, according to the technique to be employed: (I) resin infiltration (II) 30% diamine silver fluoride, (III) just daily flossing by the patient. All subjects will receive placebo treatments performed in other groups. The teeth will be evaluated by clinical and radiographic exams at baseline and after 1, 3, 6, 12, 18 and 24 months. In 1, 3 and 18 months will just be evaluated aspects related to the biofilm.

ELIGIBILITY:
Inclusion Criteria:

* Primary teeth: distal surface of the first molar, mesial surface of the second molar and distal surface of the second molar (when the first permanent molar is present) with initial caries lesion (ICDAS 1, 2 or 3).
* Permanent teeth: distal surface of the first premolar, mesial surface of the second premolar, distal surface of the second premolar, mesial surface of the first molar, distal surface of the first molar and mesial surface of the second molar with initial caries lesion (ICDAS 1, 2 or 3).

Exclusion Criteria:

* Mesial surface of the first primary molar/premolar by the smaller contact with the distal surface of the canines. It will be also excluded the surfaces that show proximal restorations, sealants, cavities, defects, as well as intact teeth.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 183 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
progression of initial lesion caries | 12 and 24 months

SECONDARY OUTCOMES:
approximal plaque reduction | 1, 3, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Braga MM, Mendes FM, De Benedetto MS, Imparato JC. Effect of silver diammine fluoride on incipient caries lesions in erupting permanent first molars: a pilot study. J Dent Child (Chic). 2009a;76(1):28-33. Braga MM, Morais CC, Nakama RC, Leamari VM, Siqueira WL, Mendes FM. In vitro performance of methods of approximal caries detection in primary molars. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009b;108(4):e35-41. Cagetti MG, Campus G, Sale S, Cocco F, Strohmenger L, Lingström P. Association between interdental plaque acidogenicity and caries risk at surface level: a cross sectional study in primary dentition. Int J Paediatr Dent. 2011;21(2):119-25. Ekstrand KR, Bakhshandeh A, Martignon S. Treatment of proximal superficial caries lesions on primary molar teeth with resin infiltration and fluoride varnish versus fluoride varnish only: efficacy after 1 year. Caries Res. 2010;44(1):41-6.
- [Derived] Mattos-Silveira J, Floriano I, Ferreira FR, Vigano ME, Frizzo MA, Reyes A, Novaes TF, Moriyama CM, Raggio DP, Imparato JC, Mendes FM, Braga MM. New proposal of silver diamine fluoride use in arresting approximal caries: study protocol for a randomized controlled trial. Trials. 2014 Nov 19;15:448. doi: 10.1186/1745-6215-15-448. PMID 25409545